CLINICAL TRIAL: NCT03320291
Title: Long-term Evaluation of Primary Trapeziectomy and Placement of a RegJoint Implant in the Treatment of Rhizarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Socorro ORTIZ, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-Regjoint_TMC
Record Dates: First submitted 2017-10-10; First posted 2017-10-25 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Rhizarthrosis
Keywords: Rhizarthrosis; Regjoint; Trapeziectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regjoint (Experimental)
  Interventions: Device: Regjoint

INTERVENTIONS:
Device: Regjoint — Implant of poly-L / D-lactide (Regjoints®) in the treatment of trapezo-metacarpal osteoarthritis

SUMMARY:
In a society based on the use of everyday tools and objects, the loss of function of one or both thumbs due to Rhizarthrosis can drastically reduce the quality of life. Many patients are refractory to preservative treatments.Therefore, multiple arthroplasty techniques were developed.

Trapeziectomy, with or without tendon interposition, gives very good results in terms of pain, function or force. However, it can result in a reduction of the size of the column of the thumb, therefore leading to a loss of force.

Replacement of the trapezo-metacarpal joint with prosthetic material is also proposed and has the advantage to avoid the reduction of the thumb column. Several models are available, mono or bipolar, with a conical or hemispherical cup. Another option is the placement of implants. They were first used when a partial trapeziectomy was possible to counter the collapse of the column and are made of different materials such as metal, silicone, ceramic, pyrocarbon , and gelfoam.

The bioabsorbable poly-LD-lactide implant (PLDLA) is a relatively new possibility for the reconstruction of small joints. Studies have previously revealed that the PLDLA implant is biocompatible and represents a good alternative to arthroplasty by tendon interposition in the reconstruction of the trapezo-metacarpal articulation with osteoarthritis.

In this study, the investigators will investigate the long term effects (1 year after placement) of the Regjoint, a poly-LD-lactide implant (PLDLA).

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years
* Patients having had a trapeziectomy for more than one year, because of chronic Rhizarthrosis defined by pain and Radiographic Signs, aka articular pinching, bone erosion and potential subluxation of the trapezo-metacarpal joint.

Exclusion Criteria:

* Surgery less than 1 year ago.
* Concomitant pathology of the thumb or wrist (Recent injury or trauma, Quervain tenosynovitis, Carpal tunnel syndrome, Dupuytren, jumping finger).
* Trapeziectomy secondary to distal prosthesis and scaphoidectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Pain visual assessment scale (EVA scale) | 1 year post surgery
  Pain evaluation in the thumb column by means of the EVA scale. The EVA scale consists of a 10cm graduated strip. The patient must point its pain level on the strip: 0 cm means 'no pain' (one end of the strip) and 10 cm means 'unbearable pain' (other end of the strip).
Quick-DASH questionnaire | 1 year post surgery
  Evaluation of the return to daily life activities (work and sport)
Prehension force | 1 year post surgery
  Measured with a Standard Dynamometer or Hydraulic Pinch Gauge, with the contralateral hand used for comparison.
Maximal amplitude of the articulation | 1 year post surgery
  Measurement of the angle between the axis of the thumb and the index finger, palmar, with a goniometer
Maximal amplitude of the articulation | 1 year post surgery
  Measurement of the angle between the axis of the thumb and the index finger, radial, with a goniometer
Eroded depth | 1 year post surgery
  Evaluation of the bone erosion by means of a radiography (face/profile/oblique). Measure of the degree of subluxation/dislocation.
Kapandji score | 1 year post surgery
  Evaluation of the mobility of the thumb carpal-metacarpal joint
metacarpus length | 1 year post surgery
  Computed by radiography
metacarpal space length | 1 year post surgery
  Computed by radiography

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Gason, MD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - Clinique du Parc Léopold, Brussels

IPD SHARING:
Plan to Share IPD: No